CLINICAL TRIAL: NCT01788072
Title: INtranasal OXyTocin for the Treatment of Autism Spectrum Disorders (ASD)
Brief Title: INtranasal OXyTocin for the Treatment of Autism Spectrum Disorders
Acronym: INOXT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: McMaster University (Other); Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INOXT-10-2013
Record Dates: First submitted 2013-02-07; First posted 2013-02-11 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2018-01

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism Spectrum Disorders; Oxytocin; Adults
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Oxytocin (Active Comparator)
  Interventions: Drug: Intranasal Oxytocin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Intranasal Oxytocin — 24 IU taken twice daily (BID), in the morning and at noon/early afternoon
  Other Names: Syntocinon
  Arms: Intranasal Oxytocin
Drug: Placebo — 24 IU taken twice daily (BID), in the morning and at noon/early afternoon
  Arms: Placebo

SUMMARY:
There is substantial evidence from animal model and healthy control data, that oxytocin is involved in the modulation of social cognition. In addition, recent genetics and plasma level studies suggest a possible role for oxytocin in the pathophysiology of Autism Spectrum Disorders (ASD). As a large number of children with ASD are transitioning into adulthood and will likely require treatment, the lack of data to make meaningful treatment recommendations to facilitate adult living is an urgent issue. This study will examine the effect of intranasal oxytocin (IN-OXT) on social function in adults with ASD. It is hypothesized that IN-OXT will be superior to placebo in improving social function by the end of study treatment.

ELIGIBILITY:
Inclusion Criteria

1. Male or female outpatients 18-45 years of age, inclusive
2. Meet Diagnostic and Statistical Manual of Mental Disorders. Diagnostic and Statistical Manual (DSM-V) criteria will be established by a clinician with expertise with individuals with ASD. Best estimate Diagnosis will be reached using DSM-V criteria, the Autism Diagnostic Observation Schedule (ADOS) and the Autism Diagnostic Interview (ADI-R).
3. Have a Clinical Global Impression-Severity (CGI-S) score ≥ 4 (moderately ill) at Screening.
4. Verbal scale Intelligence Quotient (IQ) ≥ 70
5. If already receiving stable concomitant medications affecting behavior, have stable regimens with no changes during the preceding 1 month prior to Screening (with the exception of fluoxetine, where a period of 6 weeks is needed), and will not electively initiate new or modify ongoing medications for the duration of the study
6. If already receiving stable non-pharmacological educational, behavioral, and/or dietary interventions, have continuous participation during the preceding 3 months prior to Screening, and not electively initiate new or modify ongoing interventions for the duration of the study
7. Have normal physical examination and laboratory test results at screening. If abnormal, the finding(s) must be deemed clinically insignificant by the Treating Clinician.
8. Ability to speak and understand English sufficiently to allow for the completion of all study assessments
9. Ability to obtain written informed consent from the subject (if developmentally appropriate), or ability to obtain written informed consent from their surrogate decision maker (SDM), if the subject is unable to provide consent.

Exclusion Criteria

1. Patients born prior to 28 weeks gestational age
2. Patients with a primary psychiatric diagnosis other than ASD
3. Patients with a medical history of neurological disease, including, but not limited to, epilepsy/seizure disorder, movement disorder, tuberous sclerosis, fragile X, and any other known genetic syndromes, or known abnormal brain MRI/structural lesion. Exceptions: 1) simple febrile seizures, 2) epilepsy/ seizure free for at least 2 years prior to Screening
4. Pregnant female patients, sexually active female patients on hormonal birth control and sexually active females who do not use at least two types of non-hormonal birth control
5. Patients with evidence or history of malignancy or any significant hematological, endocrine, cardiovascular (including any rhythm disorder), respiratory, renal, hepatic, or gastrointestinal disease
6. Patients with one or more of the following: HIV, Hepatitis B virus, Hepatitis C virus, hemophilia (bleeding problems, recent nose and brain injuries), abnormal blood pressure (hypotension or hypertension), drug abuse, immunity disorder or severe depression.
7. Patients unable to tolerate venipuncture procedures for blood sampling
8. Patients who are currently taking oxytocin or have taken intranasal oxytocin in the past with no response
9. Patients with a sensitivity to oxytocin or any components of its formulation

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Efficacy of intranasal oxytocin vs. placebo on social function in adults with ASD | 12 weeks
  This will be measured by the Clinical Global Impressions - Improvement Scale - Social (CGI-I-Social).

SECONDARY OUTCOMES:
Efficacy of intranasal oxytocin vs. placebo on a continuous measure of social cognition in adults with ASD | 12 weeks
  This will be measured by the Revised Eyes Test
Efficacy of intranasal oxytocin vs. placebo on a continuous measure of social function in adults with ASD | 12 weeks
  This will be measured by the Vineland Adaptive Behavior Scale (VABS-II)
Efficacy of intranasal oxytocin vs. placebo on a continuous measure of social responsiveness in adults with ASD | 12 weeks
  This will be measured by the Social Responsiveness Scale (SRS-2)
Efficacy of intranasal oxytocin vs. placebo on a continuous measure of social responsiveness in adults with ASD | 12 weeks
  This will be measured by the Aberrant Behavior Checklist (ABC)
Safety and tolerability of intranasal oxytocin in adults with ASD | 12 weeks
  This will be measured by the Safety Monitoring Uniform Report Form (SMURF)
Safety and tolerability of intranasal oxytocin in adults with ASD | 12 weeks
  This will be measured by the Clinical Global Impressions - Improvement Scale - Global (CGI-I-Global)
Efficacy of intranasal oxytocin vs. placebo on quality of life | 12 weeks
  This will be measured by the World Health Organization Quality of Life Survey (WHOQOL-BREF)
Efficacy of intranasal oxytocin vs. placebo on anxiety | 12 weeks
  This will be measured by the Symptom Checklist 90-Revised (SCL-90-R)

CONTACTS AND LOCATIONS:
Overall Officials: Evdokia Anagnostou, M.D., Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital; Marc Woodbury-Smith, M.D., Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton, Hamilton, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No